CLINICAL TRIAL: NCT04665414
Title: Value of Transvaginal Ultrasound, Transvaginal Sonographic Elastography and MRI for the Diagnosis of Adenomyosis
Brief Title: Diagnosis of Adenomyosis Using Ultrasound, Elastography and MRI
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Dr. med. Sebastian Daniel Schäfer, Head of Gynecology, University Hospital Muenster
Other Study IDs: Schäfer_Adenomyosis
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Endometriosis; Adenomyosis
Keywords: adenomyosis; endometriosis; MRI; elastography; ultrasound; hysterectomy
MeSH Terms: conditions — Endometriosis; Adenomyosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — preoperative MRI
Diagnostic Test: transvaginal ultrasound — preoperative transvaginal ultrasound
Diagnostic Test: transvaginal ultrasound elastography — preoperative transvaginal ultrasound elastography

SUMMARY:
comparison of transvaginal ultrasound, transvaginal ultrasound elastography and MRI for the diagnosis of adenomyosis in patients receiving hysterectomy afterwards

ELIGIBILITY:
Inclusion Criteria:

* dysmenorrhea
* dyspareunia
* non cyclic lower abdominal pain
* hypermenorrhea
* menometrorrhaghia
* pain while compressing the Uterus during gyn exam
* Patient wants to participate
* Patient will receive hysterectomy

Exclusion Criteria:

* Patient declines to participate
* contraindications against MRI
* contraindications against ultrasound
* minor
* cannot give informed consent
* no hysterectomy planned

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: all patients in accordance with eligibility criteria registered to receive hysterectomy because of a suspicion of adenomyosis according to the above criteria
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
sensitivity MRI | through study completion, an average of 1 year
  sensitivity MRI
specificity MRI | through study completion, an average of 1 year
  specificity MRI
sensitivity transvaginal ultrasound | through study completion, an average of 1 year
  sensitivity transvaginal ultrasound
specificity transvaginal ultrasound | through study completion, an average of 1 year
  specificity transvaginal ultrasound
sensitivity transvaginal ultrasound elastography | through study completion, an average of 1 year
  sensitivity transvaginal ultrasound elastography
specificity transvaginal ultrasound elastography | through study completion, an average of 1 year
  specificity transvaginal ultrasound elastography
sensitivity intraoperative ENZIAN FA | through study completion, an average of 1 year
  sensitivity intraoperative ENZIAN FA
specificity intraoperative ENZIAN FA | through study completion, an average of 1 year
  specificity intraoperative ENZIAN FA

SECONDARY OUTCOMES:
sensitivity and specificity of single sonographic or MRI criteria or combinations thereof | through study completion, an average of 1 year
  sensitivity and specificity of single sonographic or MRI criteria or combinations thereof

CONTACTS AND LOCATIONS:
Overall Officials: se D Schaefer, MD PhD, Principal Investigator — University Hospital Muenster, Germany
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
data will be shared upon reasonable request according to regulations